CLINICAL TRIAL: NCT02303951
Title: Neoadjuvant Treatment With the Combination of Vemurafenib, Cobimetinib and Atezolizumab in Limited Metastasis of Malignant Melanoma (AJCC Stage IIIC/IV) and Integrated Biomarker Study: a Single Armed, Two Cohort, Phase II EADO Trial NEO-VC
Brief Title: Neoadjuvant Vemurafenib + Cobimetinib + Atezolizumab in Melanoma: NEO-VC
Acronym: NEO-VC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The main reason for the early termination is the low recruitment rate.
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EADO_VC_NEO_1
Record Dates: First submitted 2014-11-13; First posted 2014-12-01 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2020-05

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — Vemurafenib; cobimetinib; atezolizumab

STUDY DESIGN:
Intervention Model Description: Single armed, two-cohort Cohort I: Treatment with cobimetinib + vemurafenib; 45 patients enrolled; recruitment closed Cohort II: Treatment with cobimetinib + vemurafenib + atezolizumab; 45 patients planned; recruitment open
Oversight: Data Monitoring Committee: No

ARMS (1):
- vemurafenib + cobimetinib + atezolizumab (Experimental): Run-In (week 1-4):
  * Day 1-21: vemurafenib 960 mg bid orally + cobimetinib 60 mg od orally
  * Day 22-28: vemurafenib 720 mg bid orally
  Triple-Treatment (week 5 ongoing):
  atezolizumab 840 mg Q2W i.v. + vemurafenib 720 mg bid orally + cobimetinib 60 mg od 21/7 orally (vemurafenib: daily intake; cobimetinib: 3 weeks on drug, 1 week off)
  Interventions: Drug: Vemurafenib; Drug: Cobimetinib; Drug: Atezolizumab

INTERVENTIONS:
Drug: Vemurafenib — Run-In: Day 1-21 960 mg bid orally, Day 22-28 720 mg bid orally Triple-Treatment (week 5 ongoing): 720 mg bid orally
  Other Names: Zelboraf
Drug: Cobimetinib — Run-In: Day 1-21 60 mg od orally Triple-Treatment (week 5 ongoing): 60 mg od 21/7 orally (3 weeks on drug, 1 week off)
  Other Names: Cotellic
Drug: Atezolizumab — Triple-Treatment (week 5 ongoing): 840 mg Q2W i.v
  Other Names: Tecentriq

SUMMARY:
Evaluation of the efficacy, safety and biologic effects of neo-adjuvant treatment with vemurafenib + cobimetinib + atezolizumab in patients with limited metastasis of melanoma in stage IIIC/IV melanoma.

DETAILED DESCRIPTION:
Patients with hardly resectable/unresectable limited metastasis in malignant melanoma stages IIIC/IV (AJCC 2010) carrying the BRAF V600 mutation, in order to achieve operability are enrolled in the NEO-VC-study. The main aim of this study is to achieve operability in a higher percentage of patients by neoadjuvant treatment through shrinkage of the tumors. Patients with operable stage IV disease show an impressive survival benefit with long term (5 y.) survival rates around 30 %. Only a percentage of up to 20 % can presently be treated by complete metastasectomy. This percentage may be enlarged by pre-treatment with an efficacious antitumor drug.

ELIGIBILITY:
Inclusion Criteria:

1. Signed ICF
2. Age ≥ 18 years
3. Histologically confirmed Stage IV (metastatic) or unresectable Stage IIIC (locally advanced) melanoma, as defined by the AJCC, 7th revised edition

   1. Naïve to prior systemic anti-cancer therapy for melanoma, with the following exceptions: Adjuvant treatment with IFN, IL-2, or vaccine therapies, if discontinued at least 28 days prior to initiation of study treatment
   2. Adjuvant treatment with herbal therapies, if discontinued at least 7 days prior to initiation of study treatment
4. Documentation of BRAFV600 mutation-positive status in melanoma tumor tissue (archival or newly obtained) through use of a clinical mutation test approved by the local health authority
5. ECOG of 0 or 1
6. Decision of eligibility for neoadjuvant combined vem+cobi+atezo treatment by in-terdisciplinary tumor board. Patient with limited numbers of metastases and few organ systems involved should be selected, making surgical resection after neo-adjuvant treatment probable.
7. Measurable disease by RECIST V1.1 criteria (must be outside the CNS)
8. Adequate hematologic and end-organ function, defined by the following laboratory test results, obtained within 14 days prior to initiation of study treatment, with the exception of amylase, lipase, and LDH where up to 28 days is acceptable

   * ANC ≥ 1.5 × 109/L without granulocyte colony-stimulating factor support
   * WBC count ≥ 2.5 × 109/L
   * Lymphocyte count ≥ 0.5 × 109/L
   * Platelet count ≥ 100 × 109/L without transfusion
   * Hemoglobin ≥ 9 g/dL without transfusion
   * Serum albumin ≥ 2.5 g/dL
   * Total bilirubin ≤ 1.5 × ULN
   * AST and ALT ≤ 2.0 x ULN
   * Amylase and lipase ≤ 1.5 x ULN
   * ALP ≤ 2.5 × ULN or, for patients with documented liver or bone metastases, ALP ≤ 5 × ULN
   * Serum creatinine ≤ 1.5 × ULN or CrCl ≥ 40mL/min on the basis of measured CrCl from a 24-hour urine collection or Crockcroft-Gault glomerular filtration rate estimation:
   * CrCL= ((140-age) x (weight in kg) x (72 x (serum creatinine in mg/dL)-1) (x 0.85 if female)
   * For patients not receiving therapeutic anticoagulation: INR or aPTT ≤ 1.5 × ULN within 28 days prior to initiation of study treatment
   * For patients receiving therapeutic anticoagulation: stable anticoagulant regi-men and stable INR during the 28 days immediately preceding initiation of study treatment
9. For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as defined below:

   1. With female partners of childbearing potential, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for at least 6 months after the last dose of study treatment. Men must refrain from donating sperm during this same period.
   2. With pregnant female partners, men must remain abstinent or use a condom during the treatment period and for 6 months after the last dose of study treatment to avoid exposing the embryo.
   3. The reliability of sexual abstinence should be evaluated in relation to the dura-tion of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence and withdrawal are not acceptable methods of contraception
10. For WOCBP: agreement to remain abstinent (refrain from heterosexual inter-course) or use a contraceptive method with a failure rate of <1% per year during the treatment period and for 6 months after the last dose of study treatment

    1. A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state, and has not undergone surgical sterilization
    2. Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices (IUD), and copper IUDs.
    3. Hormonal contraceptive methods must be supplemented by a barrier method. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence and withdrawal are not acceptable methods of contraception.
11. Female subjects who are lactating have to discontinue nursing prior to the first dose of study drug and must refrain from nursing throughout the treatment period and for 14 days following the last dose of study drug.

Exclusion Criteria:

1. Candidates for direct surgery: patients with single site easily resectable metasta-sis
2. Major surgical procedure or significant traumatic injury within 2 weeks prior to first dose of study drug treatment
3. Palliative radiotherapy within 14 days prior to initiation of study treatment
4. Active malignancy (other than BRAFV600 mutation-positive melanoma) or malig-nancy within 3 years prior to screening are excluded, with the exception of resected melanoma, resected BCC, resected cuSCC, resected carcinoma in situ of the cervix, resected carcinoma in situ of the breast, in situ prostate cancer, limited-stage bladder cancer, or any other curatively treated malignancies from which the patient has been disease-free for at least 3 years

   a. Patients with a history of isolated elevation in prostate-specific antigen in the absence of radiographic evidence of metastatic prostate cancer are eligible for the study.
5. A history of or evidence of retinal pathology on ophthalmologic examination that is considered a risk factor for neurosensory retinal detachment, CSCR, RVO, or ne-ovascular macular degeneration

   a. Patients will be excluded from study participation if they currently are known to have any of the following risk factors for RVO: i. History of serous retinopathy ii. History of RVO iii. Evidence of ongoing serous retinopathy or RVO at baseline
6. History of clinically significant cardiac dysfunction, including the following:

   1. Poorly controlled hypertension, defined as sustained, uncontrolled, non-episodic baseline hypertension consistently above 159/99mmHg despite opti-mal medical management
   2. Unstable angina, or new-onset angina within 3 months prior to initiation of study treatment
   3. Symptomatic congestive heart failure, defined as NYHA Class II or higher
   4. Myocardial infarction within 3 months prior to initiation of study treatment
   5. Unstable arrhythmia
   6. History of congenital long QT syndrome
   7. QTcF ≥480 ms at screening, or uncorrectable abnormalities in serum electro-lytes
   8. LVEF below the institutional lower limit of normal or below 50%, whichever is lower
7. Untreated or actively progressing CNS lesions (carcinomatous meningitis)
8. Patients with a history of CNS lesions are eligible, provided that all of the following criteria are met:

   1. Measurable disease, per RECIST v1.1, must be present outside the CNS
   2. All known CNS lesions have been treated with radiotherapy or surgery
   3. CNS lesions have not been treated with whole-brain radiotherapy, except in patients who underwent definitive resection of or stereotactic therapy for all radiologically detectable parenchymal brain lesions
   4. Absence of interim progression must be confirmed by radiographic study within 4 weeks prior to initiation of study treatment. If new CNS metastases are suspected during the screening period, a confirmatory radiographic study is required prior to initiation of study treatment
   5. Any radiotherapy or surgery must be completed ≥ 4 weeks prior to initiation of study treatment
   6. There is no ongoing requirement for corticosteroids, and any prior corticosteroid treatment must be discontinued ≥ 2 weeks prior to initiation of study treatment. Treatment with an anticonvulsant at a stable dose is allowed
   7. No history of intracranial hemorrhage from CNS lesions
9. History of metastases to brain stem, midbrain, pons, or medulla, or within 10 mm of the optic apparatus
10. History of leptomeningeal metastatic disease
11. Anticipated use of any concomitant medication during or within 7 days prior to initiation of study treatment that is known to cause QT prolongation. Patients with regular amiodaron intake in the last 365 days cannot be included.
12. Uncontrolled diabetes or symptomatic hyperglycemia
13. History of malabsorption or other clinically significant metabolic dysfunction that may interfere with absorption of oral study treatment
14. Pregnancy or lactation period or intention to become pregnant during the study.

    a. WOCBP must have a negative serum pregnancy test result within 7 days prior to initiation of study treatment
15. Prior allogeneic stem cell or solid organ transplantation
16. History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan

    a. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
17. Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus ery-thematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions:

    a. Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid-replacement hormone may be eligible for the study after discussion with and approval by the Medical Monitor b. Patients with controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible for the study after discussion with and approval by the Medical Monitor c. Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with der-matologic manifestations only are eligible for the study provided all of following conditions are met: i. Rash must cover < 10% of body surface area ii. Disease is well controlled at baseline and requires only low-potency topical corticosteroids iii. No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral cor-ticosteroids within the previous 12 months
18. Known clinically significant liver disease, including alcoholism, cirrhosis, fatty liver, and other inherited liver disease as well as active viral disease including:

    1. Positive HIV test at screening
    2. Active HBV infection, defined as having a positive HBsAg test at screening Patients with a past or resolved HBV infection, defined as having a negative HBsAg test and a positive total HBcAb test at screening, are eligible for the study
    3. Active HCV infection, defined as having a positive HCV antibody test and a positive HCV RNA test at screening
19. Active tuberculosis
20. Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
21. Any Grade ≥ 3 hemorrhage or bleeding event within 4 weeks prior to initiation of study treatment
22. History of stroke, reversible ischemic neurological defect, or transient ischemic at-tack within 6 months prior to initiation of study treatment
23. Current severe, uncontrolled systemic disease or any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or could jeopardize the safety of the patient and their compliance in the study
24. Signs or symptoms of clinically relevant infection and/or treatment with therapeutic systemic antibiotics within 2 weeks prior to initiation of study treatment

    a. Patients receiving prophylactic antibiotics are eligible for the study
25. Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during the course of the study
26. Treatment with systemic immunosuppressive medication within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during the study

    1. Patients who have received acute, low-dose systemic immunosuppressant medication ≥ 4 weeks prior to ini-tiation of study treatment or a one-time pulse dose of systemic immunosup-pressant medication are eligible for the study.
    2. The use of inhaled corticosteroids for chronic obstructive pulmonary disease or asthma, mineralocorticoids , or low-dose corticosteroids for patients with orthostatic hypotension or adrenocortical insufficiency is allowed.
27. Known hypersensitivity to biopharmaceutical agents produced in Chinese hamster ovary cells
28. Known hypersensitivity to any component of the atezo, cobi, or vem formulations
29. History of severe allergic, anaphylactic or other hypersensitivity reactions to chi-meric or humanized antibodies or fusion proteins
30. Treatment with any other investigational agent or participation in another clinical study with therapeutic intent within 4 weeks of the start of study treatment.
31. Inability or unwillingness to swallow pills
32. Any psychological, familial, sociological, or geographical conditions that may hamper compliance with the protocol and follow-up after treatment discontinuation
33. Requirement for concomitant therapy or food that is prohibited during the study, as described in Sections 10.10 and 10.11.
34. Patient is unable to comply with the study protocol for any other reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-01-22 (Actual); Primary Completion 2020-05-14 (Actual); Study Completion 2020-05-14 (Actual)

PRIMARY OUTCOMES:
Percent of patients who actually become resectable and are resected | Following 18 weeks of combined treatment
  Percentage of patients becoming operable after the combined treatment within 18 weeks. The primary research question is the difference of this observed proportion with verum-treatment in the study which is compared to an assumed/known proportion without treatment based on an estimation of the scientific community

SECONDARY OUTCOMES:
Progression free survival time after resection | Following 18 weeks of combined treatment
  Progression free survival time after resection, in the group who actually underwent complete resection
Progression free survival | Following 6 and 12 months of combined treatment
  Progression free survival rates at 6 and 12 months after start of treatment
Objective response | Up to 29 months
  Rate of objective responses
Tolerability (Number of patients with adverse events and number of patients who prematurely discontinued treatment due to adverse events) | Up to 29 months
  Number of patients with adverse events and number of patients who prematurely discontinued treatment due to adverse events
Overall survival | Up to 29 months
  Overall survival in the total study population
Progression free survival time | Up to 29 months
  Progression free survival time in the total study population

OTHER OUTCOMES:
Detection of biomarkers for response to vemurafenib + cobimetinib + atezolizumab in metastatic tumor tissue | Screening (= pre-treatment) and following 18 weeks of combined treatment
  Detection of biomarkers for response to vemurafenib + cobimetinib + atezolizumab by analysis of baseline metastatic tumor tissue and comparing metastatic tumor tissues pretreatment and post treatment:
  * Changes in key cell signaling pathway in immunohistochemistry (IHC)
  * Changes in T-cell infiltration and expression of immune-modulators by IHC (Immunohistochemistry)
Detection of biomarkers for response to vemurafenib + cobimetinib in blood samples | Screening (= pre-treatment)
  Detection of biomarkers for response to vemurafenib + cobimetinib by analysis of baseline blood samples:
  * Changes in key cell signaling pathway in immunohistochemistry (IHC)
  * Changes in T-cell infiltration and expression of immune-modulators by IHC
Detection of differences in gene expression in metastatic tumor tissue | Screening (pre-treatment) and following 18 weeks of combined treatment
  Differences in gene expression, oncogenic mutation/copy number alteration profiles, and oncogenic signaling pathway status by analysis of baseline metastatic tumor tissue and comparing metastatic tumor tissues pretreatment and post treatment:
  * Changes in oncogenic mutation profiles by whole exome sequencing (WES)
  * Changes in transcriptome profiles by RNAseq
Detection of differences in gene expression in blood samples | Screening (pre-treatment)
  Differences in gene expression, oncogenic mutation/copy number alteration profiles, and oncogenic signaling pathway status by analysis of baseline blood samples:
  * Changes in oncogenic mutation profiles by whole exome sequencing (WES)
  * Changes in transcriptome profiles by RNAseq

CONTACTS AND LOCATIONS:
Overall Officials: Claus Garbe, Prof., Principal Investigator — University Hospital Tübingen
Locations (7):
- France (3):
  - Department of Dermatology & Skin Cancer University Hospital La Timone, Aix-Marseille University, Marseille
  - Department of Dermatology, University Hospital of Nantes, Nantes
  - Hopital Saint-Louis Hopitaux Universitaires Saint-Louis Laboisiere Fernand-Widal, Paris
- Germany (4):
  - Department of Dermatology, Elbe Hospital, Buxtehude
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Department of Dermatology, University Hospital, Kiel
  - University hospital Tübingen, Tübingen

REFERENCES:
- [Derived] Gorry C, McCullagh L, O'Donnell H, Barrett S, Schmitz S, Barry M, Curtin K, Beausang E, Barry R, Coyne I. Neoadjuvant treatment for stage III and IV cutaneous melanoma. Cochrane Database Syst Rev. 2023 Jan 17;1(1):CD012974. doi: 10.1002/14651858.CD012974.pub2. PMID 36648215